CLINICAL TRIAL: NCT03547947
Title: Clinical and Radiological Outcomes of Medacta Shoulder System
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P06.001.01
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Rotator Cuff Tear Arthropathy; Rheumatoid Arthritis Shoulder; Avascular Necrosis; Fracture; Revision of Shoulder Arthroplasty
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Osteonecrosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Medacta Shoulder System — Total Shoulder Arthroplasty

SUMMARY:
This is a post-marketing surveillance on Medacta Shoulder System

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patient with one of the following diagnosis:

Primary osteoarthritis Secondary osteoarthritis Cuff tear arthropathy; insufficient rotator cuff Acute fracture (<21d) Rheumatoid or inflammatory arthritis Avascular necrosis Other posttraumatic condition Revision of shoulder arthroplasty

Exclusion Criteria:

* Patients with malignant diseases (at the time of surgery)
* Patients with proven or suspect infections (at the time of surgery)
* Patients with functional deficits other than dysfunction of the shoulder (at the time of surgery)
* Patients with known incompatibility or allergy to products materials (at the time of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring TSA and who are suitable to receive Medacta Shoulder System will be proposed to take part to the current post-marketing surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2031-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Clinical outcome | 1, 2, 5 and 10 years
  Constant & Murley Score
Functional outcome | 1, 2, 5 and 10 years
  Oxford Shoulder Score
Radiographic performance of the implants | 3 months, 1, 2, 5 and 10 years
  presence of radiolucencies
Quality of life | 1, 2, 5 and 10 years
  EQ-5D
Adverse events | up to 10 years
  record of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Zumstein, Prof Dr. Med, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (6):
- Clinique du Sport et de Chirurgie Orthopédique, Marcq-en-Barœul, France
- Klinik und Poliklinik für Orthopädie, Physikalische Medizin und Rehabilitation, München, Germany
- Switzerland (4):
  - Orthopädie Sonnenhof, Bern, Canton of Bern
  - Inselspital, Bern
  - Lindenhofspital, Bern
  - Klinik für Orthopädische Chirurgie und Traumatologie des Bewegungsapparates, Kantonsspital St.Gallen,, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No